CLINICAL TRIAL: NCT00055861
Title: PHASE 2 STUDY OF BEVACIZUMAB IN COMBINATION WITH DOCETAXEL IN PATIENTS WITH ADVANCED BREAST CANCER
Brief Title: Bevacizumab and Docetaxel in Treating Women With Locally Advanced or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01433; OSU 0218; NCI-2715; OSU-0218; UCHSC-01239; CDR0000271359
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Recurrent Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Docetaxel

ARMS (1):
- Treatment (bevacizumab, docetaxel) (Experimental): Patients receive bevacizumab IV over 30-90 minutes on weeks 1 and 3 and docetaxel IV over 60 minutes on weeks 1, 2, and 3. Treatment repeats every 4 weeks for up to 12 courses in the absence of unacceptable toxicity or disease progression.
  Interventions: Biological: bevacizumab; Drug: docetaxel; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Drug: docetaxel — Given IV
  Other Names: RP 56976; Taxotere; TXT
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is to see if combining bevacizumab with docetaxel works in treating women who have locally advanced or metastatic breast cancer. Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies, such as bevacizumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or deliver cancer-killing substances to them. Combining chemotherapy with monoclonal antibody therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the response rate in women with locally advanced or metastatic breast cancer treated with bevacizumab and docetaxel.

II. Determine the side effects of this regimen in these patients. III. Correlate soluble activated endothelial cell markers and adhesion molecules, quantitation of tumor and/or endothelial cell apoptosis, and quantitation of microvessel density with clinical outcome in patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients receive bevacizumab IV over 30-90 minutes on weeks 1 and 3 and docetaxel IV over 60 minutes on weeks 1, 2, and 3. Treatment repeats every 4 weeks for up to 12 courses in the absence of unacceptable toxicity or disease progression. After completion of 6 courses of combined treatment, patients with an ongoing response may receive bevacizumab alone in the absence of disease progression.

PROJECTED ACCRUAL: A total of 16-27 patients will be accrued for this study within 14-27 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed breast cancer

  * Local-regional recurrences or metastatic disease
* At least 1 unidimensionally measurable lesion at least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
* No history or evidence of CNS disease (e.g., primary brain tumor or any brain metastases)
* Hormone receptor status:

  * Not specified
* Female
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* More than 3 months
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* No bleeding diathesis or coagulopathy
* Bilirubin normal
* AST/ALT no greater than 2.5 times upper limit of normal
* INR less than 1.5 (patients receiving warfarin)
* Creatinine normal
* Creatinine clearance at least 60 mL/min
* No baseline proteinuria

  * Patients with proteinuria of 1+ or greater at baseline are allowed provided 24-hour urinary protein is less than 500 mg
* No symptomatic congestive heart failure
* No cardiac arrhythmia
* No uncontrolled hypertension
* No history of stroke
* No clinically significant peripheral artery disease
* No arterial thromboembolic event within the past 6 months, including any of the following:

  * Transient ischemic attack
  * Cerebrovascular accident
  * Unstable angina
  * Myocardial infarction
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No seizures not controlled with standard medical therapy
* No prior allergic reactions attributed to compounds of similar chemical or biological composition to study agents
* No psychiatric illness or social situation that would preclude study compliance
* No ongoing or active infection
* No other concurrent uncontrolled illness
* No non-healing wounds
* No significant traumatic injury within the past 28 days
* Prior adjuvant chemotherapy allowed (up to 1 regimen for metastatic disease)

  * More than 6 months since prior taxane-containing adjuvant chemotherapy
* More than 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* More than 3 weeks since prior radiotherapy
* More than 28 days since prior major surgery or open biopsy
* More than 7 days since prior fine needle aspirations other than in the breast
* More than 7 days since prior placement of a vascular access device
* No concurrent major surgical procedure
* No concurrent or recent full-dose oral or parenteral anticoagulants or thrombolytic agents (except as required to maintain patency of preexisting, permanent indwelling IV catheters)
* No other concurrent investigational agents
* No concurrent chronic daily aspirin (more than 325 mg/day) or nonsteroidal anti-inflammatory medications (known to inhibit platelet function at doses used to treat chronic inflammatory diseases)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2002-07; Primary Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Response rate according to Response Evaluation Criteria in Solid Tumors (RECIST) | Up to 4 years
  The response rate will be estimated with exact binomial 95% confidence intervals.
Side effects as assessed by the National Cancer Institute (NCI) Common Toxicity Criteria (CTC) version 2.0 | Up to 4 years

SECONDARY OUTCOMES:
Correlation of biologic studies with clinical outcomes | Up to 4 years
  Associations between laboratory endpoints (pre-study plasma VEGF and IL-8, E-selectin, P-selectin, CD31, ICAM-1, VCAM_1, CD44, PDGF, FGF, MMP-2 and MMP-9.) and response or toxicity will be investigated using Wilcoxon rank-sum tests for ordinal or continuous endpoints, or chi-square tests for binary or categorical endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Shapiro, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Ohio State University Medical Center, Columbus, Ohio